CLINICAL TRIAL: NCT05643482
Title: Hyperbaric Oxygen Therapy for Post-Concussion Syndrome: A Double-Blind, Randomized, Placebo-Controlled Pilot Study
Brief Title: Hyperbaric Oxygen Therapy for Post-Concussion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James Berry, Professor- Anesthesiology & Pain Mgmt, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2022-0697
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized between HBOT and control group with a 1:1 allocation ratio, stratified by decade of age and gender via computer generated block randomization with block size of four.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HBOT Arm (Experimental): Pressurized at 2.0 atmospheres absolute of pressure (ATA) Breathe 100% oxygen 90 minute session, 5 days per week, for 20 sessions
  Interventions: Device: Hyperbaric Oxygen Treatment
- Control Arm (Sham Comparator): Placebo Gas Pressurized at 2.0 ATA Breathe placebo gas system of 10.5% oxygen and 89.5% nitrogen to mimic the partial pressure of oxygen breathed in regular air at sea level pressure 90 minute session, 5 days per week, for 20 sessions
  Interventions: Other: Placebo gas

INTERVENTIONS:
Device: Hyperbaric Oxygen Treatment — Pressurization at 2.0 ATA with 100% oxygen
  Arms: HBOT Arm
Other: Placebo gas — Pressurization at 2.0 ATA with 10.5% oxygen to mimic normal air
  Arms: Control Arm

SUMMARY:
The purpose of this study is to decrease symptom burden, improve cognitive function, and improve quality of life outcomes in subjects with mild TBI and persisting post-concussion syndrome using Hyperbaric Oxygen Treatment compared to a sham intervention.

Specific Aims:

1. Evaluate the efficacy of hyperbaric oxygen treatment to improve outcomes for adults with persisting post-concussion syndrome. Specifically, the investigators hypothesize that a prescribed course of hyperbaric oxygen treatments (HBOT) will improve outcomes and quality of life in adults with persisting symptoms >3 months after injury.

   1. Decrease symptom burden as measured by the Rivermead Post-Concussion Symptoms Questionnaire (RPQ).
   2. Improve cognitive function as measured by the National Institutes of Health (NIH) Toolbox Cognition Battery.
   3. Improve quality of life as measured by the 36-Item Short Form Survey (SF-36).
2. Assess the safety and tolerability of hyperbaric oxygen treatments and compliance with treatment in adults with persisting post-concussion syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Must have been evaluated within 3 weeks of injury and given a diagnosis of concussion by a medical professional
* Must be experiencing persistent symptoms 3-12 months after injury as defined as having at least symptoms that are moderate to severe (score 3-4) OR at least a total score of 10 with at least 1 symptom rated moderate to severe (3-4) on the Rivermead Post-Concussion Questionnaire (RPQ).

Exclusion Criteria:

Clinically significant cardiac, neurological, psychological/psychiatric, or respiratory impairment in the opinion of the investigators, including but not limited to:

1. Pulmonary:

   * COPD with CO2 retention; previous/current imaging showing hyperinflation/air trapping/bullous disease/blebs
   * Current pneumothorax or previous spontaneous pneumothorax
2. Cardiac:

   * Uncontrolled HTN (systolic >180 or diastolic >100)
   * Known Ejection fraction < 35%
   * Pacemaker / ICD in place (not approved for chamber use)
3. Hematological/Oncological:

   * Current chemotherapeutic drug use, and past history of bleomycin use.
   * Hereditary Spherocytosis
   * Sickle cell anemia
4. Neurological and Psychological:

   * Implanted nerve stimulators
   * Uncontrolled seizure disorder
   * Drug or alcohol abuse/dependence
   * Current treatment for alcohol cessation with disulfiram
   * Claustrophobia
5. Head and Neck:

   * Inability to equilibrate the pressure of middle ears and sinuses
   * Current or previous retinal detachment
   * Retinal or vitreous surgery within the past 3 months
6. Miscellaneous:

   * Current fever or active infection
   * Implanted devices not on the approved list for use with HBOT
   * Women who are pregnant. Women with childbearing potential are required to use effective birth control if not surgically sterile or postmenopausal for >2 years.
   * Undergoing vestibular or other therapy during the intervention
   * Planning a change in medication during the intervention
7. Relative exclusion criteria: Diagnosis of the conditions listed below will require approval of the hyperbaric medicine physician for enrollment into the study.

   * Asthma
   * Optic neuritis
   * Otosclerosis surgery
   * Thoracic surgery
   * Chronic sinusitis
8. Medications: Individuals with recent (within the past six months) or concurrent use of these medications must be approved by the hyperbaric medicine physician.

   * Antabuse - Predisposes to oxygen toxicity
   * Antiseizure medications - Potential participants must have levels of their seizure medications checked within a week of their initial screening visit because low levels can predispose to oxygen toxicity. Laboratory testing must be completed by their outside treating physicians to provide to the research staff for review; the study will not obtain labs for monitoring medication levels as part of the inclusion/exclusion criteria
   * Meclizine - Predisposes to oxygen toxicity
   * Bleomycin - May cause pulmonary fibrosis that can lead to air embolism or pneumothorax in the patient receiving hyperbaric oxygen treatment.
   * Certain ointments/creams that cannot be removed - These may be allowed if covered with cotton dressings.
   * Narcotics - Can lead to cessation of the hypoxic respiratory drive.
   * Nitroprusside - HBOT vasoconstrictive effect interacts with nitroprusside's vasodilator effect, making intensive monitoring mandatory.
   * Penicillin - Predisposes to oxygen toxicity
   * Promethazine (Phenergan) - Predisposes to oxygen toxicity.
   * Corticosteroids - Decreases the threshold for oxygen toxicity.
   * Sulfamylon - Promotes CO2 buildup causing peripheral vasodilatation. When coupled with vasoconstriction, results are worse than with using either agent alone. Use silver sulfadiazine instead for wound care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Change in symptom burden as measured by the Rivermead Post-Concussion Symptoms Questionnaire-3 (RPQ-3) | Baseline, immediately after treatment
  Change in symptom burden is measured by the Rivermead Post-Concussion Symptoms Questionnaire-3 (RPQ-3) which is a 16 item questionnaire of common cognitive, behavioral, and physical symptoms experienced following a mTBI. The RPQ is rated on a 0-4 scale with scores ranging from 0-64. Higher levels of endorsement indicate more severe symptoms. The RPQ-3 is the total score of the first three items of the RPQ and includes "headaches," "feelings of dizziness," and "nausea and/or vomiting."
Change in symptom burden as measured by the Rivermead Post-Concussion Symptoms Questionnaire-3 (RPQ-3) | Baseline, 1 month after treatment
  Change in symptom burden is measured by the Rivermead Post-Concussion Symptoms Questionnaire-3 (RPQ-3) which is a 16 item questionnaire of common cognitive, behavioral, and physical symptoms experienced following a mTBI. The RPQ is rated on a 0-4 scale with scores ranging from 0-64. Higher levels of endorsement indicate more severe symptoms. The RPQ-3 is the total score of the first three items of the RPQ and includes "headaches," "feelings of dizziness," and "nausea and/or vomiting."

SECONDARY OUTCOMES:
Change in symptom burden as measured by the Rivermead Post-Concussion Symptoms Questionnaire-13 (RPQ-13) | Baseline, immediately after last treatment
  Change in symptom burden is measured by the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) which is a 16 item questionnaire of common cognitive, behavioral, and physical symptoms experienced following a mTBI. The RPQ is rated on a 0-4 scale with scores ranging from 0-64. Higher levels of endorsement indicate more severe symptoms. The RPQ-3 is the total score of the first three items of the RPQ and includes "headaches," "feelings of dizziness," and "nausea and/or vomiting." The RPQ-13 is the total score of the remaining 13 items on the RPQ scale.
Change in symptom burden as measured by the Rivermead Post-Concussion Symptoms Questionnaire-13 (RPQ-13) | Baseline, 1 month after treatment
  Change in symptom burden is measured by the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) which is a 16 item questionnaire of common cognitive, behavioral, and physical symptoms experienced following a mTBI. The RPQ is rated on a 0-4 scale with scores ranging from 0-64. Higher levels of endorsement indicate more severe symptoms. The RPQ-3 is the total score of the first three items of the RPQ and includes "headaches," "feelings of dizziness," and "nausea and/or vomiting." The RPQ-13 is the total score of the remaining 13 items on the RPQ scale.
Change in quality of life as measured by the Short Form Survey (SF-36) | Baseline, immediately after treatment
  Change in quality of life is measured by the Short Form Survey (SF-36) which consists of 36 items and measures quality of life via eight different domains including vitality, physical functioning, social functioning, emotional role, physical role, general health, social functioning, and mental health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher scores indicating better levels of function and/or better health. A positive change from Baseline indicates improvement.
Change in quality of life as measured by the Short Form Survey (SF-36) | Baseline, 1 month
  Change in quality of life is measured by the Short Form Survey (SF-36) which consists of 36 items and measures quality of life via eight different domains including vitality, physical functioning, social functioning, emotional role, physical role, general health, social functioning, and mental health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher scores indicating better levels of function and/or better health. A positive change from Baseline indicates improvement.
Global Impression of Change (GIC) | Baseline, after 5 treatment sessions (approximately 1 week after starting treatment)
  The Global Impression of Change scale is a seven-point scale in which participants are asked to rate how much the treatment has changed their activity limitations, symptoms, emotions, and overall quality of life. Possible scores range from -3 (very much worse) to +3 (very much better) with 0 being no change.
Global Impression of Change (GIC) | Baseline, after 10 treatment sessions (approximately 2 weeks after starting treatment)
  The Global Impression of Change scale is a seven-point scale in which participants are asked to rate how much the treatment has changed their activity limitations, symptoms, emotions, and overall quality of life. Possible scores range from -3 (very much worse) to +3 (very much better) with 0 being no change.
Global Impression of Change (GIC) | Baseline, after 15 treatment sessions (approximately 3 weeks after starting treatment)
  The Global Impression of Change scale is a seven-point scale in which participants are asked to rate how much the treatment has changed their activity limitations, symptoms, emotions, and overall quality of life. Possible scores range from -3 (very much worse) to +3 (very much better) with 0 being no change.
Global Impression of Change (GIC) | Baseline, after 20 treatment sessions (approximately 3 weeks after starting treatment)
  The Global Impression of Change scale is a seven-point scale in which participants are asked to rate how much the treatment has changed their activity limitations, symptoms, emotions, and overall quality of life. Possible scores range from -3 (very much worse) to +3 (very much better) with 0 being no change.
Global Impression of Change (GIC) | Baseline, 1 month post-treatment
  The Global Impression of Change scale is a seven-point scale in which participants are asked to rate how much the treatment has changed their activity limitations, symptoms, emotions, and overall quality of life. Possible scores range from -3 (very much worse) to +3 (very much better) with 0 being no change.
Percentage of participant feeling of back to normal, pre-injury self at baseline as assessed based on patient rating | Baseline
  Percentage of participant feeling of back to normal, pre-injury self at baseline is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Percent change in participant feeling of back to normal, pre-injury self as assessed based on patient rating | Baseline, after 5 treatment sessions (approximately 1 week after starting treatment)
  Percent change in participant feeling of back to normal, pre-injury self is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Percent change in participant feeling of back to normal, pre-injury self as assessed based on patient rating. | Baseline, after 10 treatment sessions (approximately 2 weeks after starting treatment)
  Percent change in participant feeling of back to normal, pre-injury self is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Percent change in participant feeling of back to normal, pre-injury self as assessed based on patient rating | Baseline, after 15 treatment sessions (approximately 3 weeks after starting treatment)
  Percent change in participant feeling of back to normal, pre-injury self is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Percent change in participant feeling of back to normal, pre-injury self as assessed based on patient rating | Baseline, after 20 treatment sessions (approximately 4 weeks after starting treatment)
  Percent change in participant feeling of back to normal, pre-injury self is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Percent change in participant feeling of back to normal, pre-injury self as assessed based on patient rating | Baseline, 1 month post-treatment
  Percent change in participant feeling of back to normal, pre-injury self is assessed based on patient rating. Participants will be asked to rate what percent they feel back to their normal, pre-injury self at baseline
Change in psychological/mood symptoms as measured by Brief Symptom Inventory (BSI) scale | Baseline, immediately after last treatment
  Change in psychological/mood symptoms is measured by Brief Symptom Inventory (BSI) scale. The Brief Symptom Inventory (BSI) (secondary outcome): contains 18 items with 3 subscales measuring Depression, Anxiety, and Somatization and total raw score represents the Global Severity Index (GSI). Scores on each of the 3 subscales range from 0-24 and total GSI scores range from 0-72. Higher scores on the subscales and total GSI are indicative of more severe psychological/mood symptoms
Change in psychological/mood symptoms as measured by Brief Symptom Inventory (BSI) scale | Baseline, 1 month after treatment
  Change in psychological/mood symptoms is measured by Brief Symptom Inventory (BSI) scale. The Brief Symptom Inventory (BSI) (secondary outcome): contains 18 items with 3 subscales measuring Depression, Anxiety, and Somatization and total raw score represents the Global Severity Index (GSI). Scores on each of the 3 subscales range from 0-24 and total GSI scores range from 0-72. Higher scores on the subscales and total GSI are indicative of more severe psychological/mood symptoms
Number of participants with adverse events | 1 month after treatment
  Safety (Tolerability) of the treatment is assessed by monitoring and evaluating Adverse events (AE)s by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for 30 days post-treatment
Number of participants who missed the treatment | 5 weeks
  The count of participants who missed the treatment is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: James Berry, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine/University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No